CLINICAL TRIAL: NCT04361253
Title: A Prospective, Randomized, Double-Masked, Placebo-Controlled Trial of High-Titer COVID-19 Convalescent Plasma (HT-CCP) for the Treatment of Hospitalized Patients With COVID-19 of Moderate Severity
Brief Title: Evaluation of SARS-CoV-2 (COVID-19) Antibody-containing Plasma thErapy
Acronym: (ESCAPE)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Futility
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kaufman, Richard Max,M.D., Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P001215
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: COVID; Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Two units of apheresis HT-CCP, collected from the same donor whenever possible, will be administered sequentially over no greater than a 24-hour period to participants randomized to Arm A. Each unit of HT-CCP will be approximately 250 mL, for a total transfused volume of approximately 500 mL.
  Interventions: Biological: High-Titer COVID-19 Convalescent Plasma (HT-CCP)
- Arm B (Placebo Comparator): Two units of FFP or FP24 (each 200-275 mL, approximately 500 mL total) will be administered sequentially to participants randomized to Arm B. (FFP/FP24 unit volumes vary more than apheresis plasma units. Two FFP/FP24 units that are approximately 250 mL apiece will be provided.)
  Interventions: Biological: Standard Plasma (FFP)

INTERVENTIONS:
Biological: High-Titer COVID-19 Convalescent Plasma (HT-CCP) — 250mL HT-CCP x2 doses given sequentially.
  Arms: Arm A
Biological: Standard Plasma (FFP) — 250mL FFP or FP24 x2 doses given sequentially.
  Arms: Arm B

SUMMARY:
In this study, investigators will determine whether the early addition of HT-CCP to standard treatment improves the clinical outcome (as assessed by the Modified WHO Ordinal Scale) of patients with COVID-19 who are hospitalized but not yet in moderate or severe ARDS.

DETAILED DESCRIPTION:
Investigators are doing this research to learn more about high-titer COVID-19 convalescent plasma (HT-CCP) transfusion as a possible treatment for people who have COVID-19, the coronavirus infection. "HT-CCP" is plasma that contains a high amount of antibodies that were made to fight off COVID-19 because it is donated by another person who has also been infected with coronavirus but has recovered, so their immune system has had enough time to make these antibodies. This study is being done to determine whether HT-CCP will help people with COVID-19 recover from their infection more quickly and lower their risk of having to go on a ventilator or reduce the time they need to stay on a ventilator. It is not yet known whether HT-CCP helps people with COVID-19, which is why the study needs to be randomized, meaning some subjects will be randomly selected to receive HT-CCP while others will be randomly selected to receive FFP.

ELIGIBILITY:
Inclusion Criteria:

1. Age >1 year.
2. Active COVID-19 infection confirmed by positive SARS-CoV-2 PCR.
3. Meets institutional criteria for admission to hospital for COVID-19.
4. Admitted to ICU or non-ICU floor within 5 days of enrollment.
5. PaO2/FiO2 >200 mmHg if intubated.
6. Patient or LAR able to provide informed consent.

Exclusion Criteria:

1. Previous treatment with convalescent plasma for COVID-19.
2. Current use of investigational antiviral therapy targeting SARS-CoV-2.
3. History of anaphylactic transfusion reaction.
4. Clinical diagnosis of acute decompensated heart failure.
5. Objection to blood transfusion.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Modified WHO Ordinal Scale (MOS) score | Day 14
  The primary outcome will be the MOS numerical score (score 0-9) where a score of 0 attributes to 'no clinical evidence of infection' and a score of 9 attributes to 'death'. The eligibility requirements for this trial select individuals at level 3 or higher on the modified scale, but the day 14 outcome can be any one of 10 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kaufman, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available upon request to the principal investigator following the publication of the primary manuscript.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months after study publication. No end date.
Access Criteria: Proposals should be submitted to rmkaufman@bwh.harvard.edu.